CLINICAL TRIAL: NCT07201363
Title: The Role of Inflammation and Fibrosis in the Development of Conduction Disorders After Transcatheter Aortic Valve Implantation
Brief Title: Biomarkers of Inflammation and Fibrosis in Conduction Disorders After TAVI
Status: Recruiting | Type: Observational
Sponsor: Clinical Hospital Center Rijeka (Other)
Collaborators: University of Rijeka, Medical Faculty (Unknown)
Responsible Party: Principal Investigator, Gordana Bacic, Principal Investigator, Clinical Hospital Center Rijeka
Other Study IDs: 003052401131
Record Dates: First submitted 2025-09-22; First posted 2025-10-01 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: TAVI(Transcatheter Aortic Valve Implantation); Conduction Disorder; Aortic Stenosis; Permanent Pacemaker Implantation
Keywords: Aortic Stenosis; Biomarkers; Conduction Disorder; Fibrosis; Inflammation; Transcatheter Aortic Valve Implantation
MeSH Terms: conditions — Arrhythmias, Cardiac; Aortic Valve Stenosis; Fibrosis; Inflammation | interventions — Echocardiography; Global Longitudinal Strain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — An additional sample od blood serum of each patient will be stored for subsequent anaysis of TGF-β1 and calprotectin. In a subpopulation of 40 patients, four specific microRNA will also be analysed from the same stored blood serum samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- The group with new-onset TAVI-related conduction disorders (CDs): The group will include patients with new-onset CD or PPI detected during the index hospitalization and a 3-month follow-up period.
  Interventions: Diagnostic Test: Biomarkers of inflammation and fibrosis in pre-procedural serum blood samples; Diagnostic Test: Transthoracic echocardiography with myocardial deformation analysis and staging according to the extent of cardiac damage related to AS
- The group without new-onset TAVI-related conduction disorders (CDs): The group will include patients without new-onset CD or PPI detected during the index hospitalization and a 3-month follow-up period.
  Interventions: Diagnostic Test: Biomarkers of inflammation and fibrosis in pre-procedural serum blood samples; Diagnostic Test: Transthoracic echocardiography with myocardial deformation analysis and staging according to the extent of cardiac damage related to AS

INTERVENTIONS:
Diagnostic Test: Biomarkers of inflammation and fibrosis in pre-procedural serum blood samples — In all patients, peripheral venous blood samples will be collected before the TAVI procedure for analysis and calculation of prespecified inflammatory and fibrosis biomarkers. In a subpopulation of 40 individuals, four specific microRNAs (miR-21, miR-29b, miR-155, and miR-146b) will be additionally analysed. The level of each biomarker will be correlated with rates of new-onset TAVI-related CDs and compared between patients with detected and patients without detected new-onset CDs.
  Other Names: C-reactive protein (CRP); Procalcitonin (PCT); Interleukin-6 (IL-6); CRP/albumin ratio (CAR); Index of Systemic Immuno-inflammation (SII); Lactate-dehydrogenase (LD); Micro ribonucleic acids (miRNAs); Ferritin; Transforming Growth Factor-β1 (TGF-β1); Calprotectin
Diagnostic Test: Transthoracic echocardiography with myocardial deformation analysis and staging according to the extent of cardiac damage related to AS — The echocardiographic stage of extravalvular cardiac damage related to AS and myocardial deformation parameters will be analysed in each patient before TAVI procedure and compared between the group with detected new-onset CDs and the group without new-onset CDs with a goal to examine their predictive value for the development of TAVI-related CDs.
  Other Names: Stage of extravalvular cardiac damage related to AS; Left ventricle global longitudinal strain (LV GLS); LV apical to basal strain ratio; Right ventricle global longitudinal strain (RV GLS); Right ventricle free wall strain (RV FWS); Myocardial work index (MWI)

SUMMARY:
Prediction of conduction disorders (CDs) in patients with severe aortic stenosis (AS) undergoing transcatheter aortic valve implantation (TAVI) is an important and complex process with a significant impact on patient outcomes. The goal of this observational prospective trial is to investigate the role of pre-procedural values of systemic biomarkers of inflammation and fibrosis in the prediction of new-onset CDs and permanent pacemaker implantation (PPI) in patients undergoing the TAVI procedure.

DETAILED DESCRIPTION:
Transcatheter aortic valve implantation (TAVI) has become an established therapeutic option for the management of severe aortic stenosis (AS) in patients at all levels of surgical risk. Significant improvements in procedural safety and efficacy, along with growing operator experience, have led to a reduction of periprocedural complications. However, the incidence of new-onset conduction disorders (CDs) remains relatively high. This represents a cause for concern, especially regarding the trend of expanding TAVI indication towards younger and lower-risk patients.

Since certain CDs and PPI after TAVI are associated with poorer outcomes, identifying patients at high risk for new-onset CDs is paramount. With careful pre-procedural planning and modification of procedural steps, it is possible to avoid the occurrence of CDs in some patients. After the procedure, more intensive and prolonged electrocardiographic (ECG) monitoring should be applied in patients at high risk. A substantial number of TAVI-related CD predictors have been identified and should be evaluated in every patient, including clinical, electrocardiographic, anatomic, and procedural-related factors.

The process of inflammation and fibrosis plays a significant role in the pathogenesis of degenerative AS, causing not only valvular changes, but also myocardial and conduction system remodeling, with limited research addressing the latter. Circulating biomarkers of inflammation and fibrosis, reflecting the underlying pathological changes of the conduction system, could potentially be correlated with the risk of TAVI-related CDs. Those biomarkers have not been investigated as predictors of the aforementioned disorders so far. Routinely and widely available inflammatory biomarkers could be used in everyday clinical practice as additional predictors for the development of TAVI-related CDs and consequently contribute to an individualized approach in planning the procedure. In accordance with certain more specific and complex biomarkers, analysis of this correlation could also contribute to understanding and clarifying the role of inflammation and fibrosis in the pathogenesis of new-onset CDs in patients undergoing the TAVI procedure.

Trial objective: To investigate the role of pre-procedural values of systemic biomarkers of inflammation and fibrosis in the prediction of new-onset CDs and permanent pacemaker implantation (PPI) in patients with severe AS undergoing TAVI procedure.

Methodology: This is an observational prospective trial that will include a minimum of 102 consecutive patients with severe AS hospitalized in Clinical Hospital Center Rijeka for a planned TAVI procedure, according to the previous Heart Team decision. In all patients, peripheral venous blood samples will be collected before the procedure for analysis and calculation of inflammatory and fibrosis biomarkers (C-reactive protein (CRP), procalcitonin (PCT), interleukin-6 (IL-6), calprotectin, lactate-dehydrogenase (LD), ferritin, CRP/albumin ratio (CAR), index of systemic immuno-inflammation (SII), and transforming growth factor-β1 (TGF- β1). In a patient subpopulation of 40 individuals, four specific microRNAs (miR-21, miR-29b, miR-155, and miR-146b) involved in the regulation of fibrosis and inflammation, will be additionally analyzed. Pre-procedural echocardiographic parameters to assess the extent of extravalvular cardiac damage related to AS and myocardial deformation analysis as a non-invasive marker of fibrosis will be evaluated and correlated with rates of new-onset TAVI-related CDs. The electrocardiogram (ECG) will be analysed before and consecutively after the procedure, during hospitalization, and at a 3-month follow-up. Patients will be assigned to a group with or without new-onset CD, whether a previously defined CD or PPI was recorded during the index hospitalization and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participate in the trial
* Diagnosis of severe AS according to current European Society of Cardiology (ESC) guidelines for valvular heart disease

Exclusion Criteria:

* Acute infectious disease
* Chronic inflammatory or autoimmune disease
* Corticosteroid or other immunosuppressive therapy
* Active malignant disease
* Liver disease accompanied by dysfunction
* Permanent pacemaker implanted previously
* An acute myocardial infarction within three months before the procedure
* A surgical procedure within three months before the procedure
* Previous surgical or transcatheter aortic valve replacement/implantation
* End-stage chronic kidney disease (eGFR <15 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The trial will include a minimum 102 consecutive patients with severe AS hospitalized in Clinical Hospital Centre Rijeka for a planned TAVI procedure, according to the previous Heart Team decision.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Pre-procedural levels of C-reactive protein (mg/L) and calprotectin (mg/L) | At hospital admission, before TAVI procedure
  The levels of C-reactive protein (mg/L) and calprotectin (mg/L) will be compared between the group with new-onset CDs and the group without new-onset CDs. The goal is to determine if their levels differ significantly between the two groups and to examine their predictive value for the development of TAVI-related CDs. For calprotectin analysis, an additional serum blood sample will be collected from every patient, and stored at -80 °C for subsequent analysis by the ELISA method.
Pre-procedural level of interleukin-6 (ng/L) | At hospital admission, before TAVI procedure
  The levels of interleukin-6 (ng/L) will be compared between the group with new-onset CDs and the group without new-onset CDs. The goal is to determine if the levels of interleukin-6 differ significantly between the two groups and to examine its predictive value for the development of TAVI-related CDs
Pre-procedural levels of procalcitonin (µg/L) and ferritin (µg/L) | At hospital admission, before TAVI procedure
  The levels of procalcitonin (µg/L) and ferritin (µg/L) will be compared between the group with new-onset CDs and the group without new-onset CDs. The goal is to determine if their levels differ significantly between the two groups and to examine their predictive value for the development of TAVI-related CDs.
Pre-procedural level of transforming growth factor-β1(pg/ml) | At hospital admission, before TAVI procedure
  The levels of transforming growth factor-β1(pg/ml) will be compared between the group with new-onset CDs and the group without new-onset CDs. The goal is to determine if the levels of TGF-β1 differ significantly between the two groups and to examine its predictive value for the development of TAVI-related CDs. For TGF-β1 analysis, an additional serum blood sample will be collected from every patient, and stored at -80 °C for subsequent analysis by the ELISA method.
Pre-procedural level of lactate-dehydrogenase (U/I) | At hospital admission, before TAVI procedure
  The levels of lactate-dehydrogenase (U/I) will be compared between the group with new-onset CDs and the group without new-onset CDs. The goal is to determine if the levels of lactate-dehydrogenase differ significantly between the two groups and to examine its predictive value for the development of TAVI-related CDs
Pre-procedural C-reactive protein to albumin ratio and index of systemic immuno-inflammation values | At hospital admission, before TAVI procedure
  The values of C-reactive protein to albumin ratio and index of systemic immuno-inflammation will be calculated and compared between the group with new-onset CDs and the group without new-onset CDs. The goal is to determine if their values differ significantly between the two groups and to examine their predictive value for the development of TAVI-related CDs.

SECONDARY OUTCOMES:
Pre-procedural levels of microRNAs (miR-21, miR-29b, miR-155, and miR-146b) in a subpopulation of 40 patients | At hospital admission, before TAVI procedure
  The levels of four microRNAs included in the regulation of the fibrosis and inflammation process will be analysed and compared between the subgroup with new-onset CDs (20 pts) and the subgroup without new-onset CDs (20 pts). A group of ten healthy individuals will be additionally included for microRNAs analysis. Serum blood samples will be collected at the time of hospitalization, before the TAVI procedure, and stored at -80 °C for subsequent analysis by polymerase chain reaction (PCR). The goal is to determine if their levels differ significantly between the two groups and analyse their correlation with other biomarkers of inflammation and fibrosis
Myocardial deformation parameters | At hospital admission, before TAVI procedure
  Left ventricle global longitudinal strain (%), right ventricle global longitudinal strain (%) and right ventricle free wall strain (%) will be compared between the group with new-onset CDs and the group without new-onset CDs, with a goal to determine if they differ significantly between the two groups and to examine their predictive value for the development of TAVI-related CDs
Left ventricle apical to basal strain ratio | At hospital admission, before TAVI procedure
  Values of the left ventricle apical to basal strain ratio will be compared between the group with new-onset CDs and the group without new-onset CDs, with a goal to determine if they differ significantly between the two groups and to examine their predictive value for the development of TAVI-related CDs
Myocardial work index (mmHg%) | At hospital admission, before TAVI procedure
  Values of myocardial work index (mmHg%) will be compared between the group with new-onset CDs and the group without new-onset CDs, with a goal to determine if they differ significantly between the two groups and to examine their predictive value for the development of TAVI-related CDs
Stage of extravalvular cardiac damage (0-4) | At hospital admission, before TAVI procedure
  Echocardiographic stages of extravalvular cardiac damage (0-4) related to AS will be compared between the group with new-onset CDs and the group without new-onset CDs, with a goal to determine if they differ significantly between the two groups and to examine their predictive value for the development of TAVI-related CDs

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital Center Rijeka, Rijeka, Croatia, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Damas F, Nguyen Trung ML, Postolache A, Petitjean H, Lempereur M, Viva T, Oury C, Dulgheru R, Lancellotti P. Cardiac Damage and Conduction Disorders after Transcatheter Aortic Valve Implantation. J Clin Med. 2024 Jan 11;13(2):409. doi: 10.3390/jcm13020409. PMID 38256543
- [Background] Ramos-Mondragon R, Galindo CA, Avila G. Role of TGF-beta on cardiac structural and electrical remodeling. Vasc Health Risk Manag. 2008;4(6):1289-300. doi: 10.2147/vhrm.s3985. PMID 19337543
- [Background] Friedman HS, Zaman Q, Haft JI, Melendez S. Assessment of atrioventricular conduction in aortic valve disease. Br Heart J. 1978 Aug;40(8):911-7. doi: 10.1136/hrt.40.8.911. PMID 687491
- [Background] Verheule S, Schotten U. Electrophysiological Consequences of Cardiac Fibrosis. Cells. 2021 Nov 18;10(11):3220. doi: 10.3390/cells10113220. PMID 34831442
- [Background] Hein S, Arnon E, Kostin S, Schonburg M, Elsasser A, Polyakova V, Bauer EP, Klovekorn WP, Schaper J. Progression from compensated hypertrophy to failure in the pressure-overloaded human heart: structural deterioration and compensatory mechanisms. Circulation. 2003 Feb 25;107(7):984-91. doi: 10.1161/01.cir.0000051865.66123.b7. PMID 12600911
- [Background] Conte M, Petraglia L, Campana P, Gerundo G, Caruso A, Grimaldi MG, Russo V, Attena E, Leosco D, Parisi V. The role of inflammation and metabolic risk factors in the pathogenesis of calcific aortic valve stenosis. Aging Clin Exp Res. 2021 Jul;33(7):1765-1770. doi: 10.1007/s40520-020-01681-2. Epub 2020 Sep 25. PMID 32978752
- [Background] Vahanian A, Beyersdorf F, Praz F, Milojevic M, Baldus S, Bauersachs J, Capodanno D, Conradi L, De Bonis M, De Paulis R, Delgado V, Freemantle N, Gilard M, Haugaa KH, Jeppsson A, Juni P, Pierard L, Prendergast BD, Sadaba JR, Tribouilloy C, Wojakowski W; ESC/EACTS Scientific Document Group. 2021 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2022 Feb 12;43(7):561-632. doi: 10.1093/eurheartj/ehab395. No abstract available. PMID 34453165
- [Background] Auffret V, Puri R, Urena M, Chamandi C, Rodriguez-Gabella T, Philippon F, Rodes-Cabau J. Conduction Disturbances After Transcatheter Aortic Valve Replacement: Current Status and Future Perspectives. Circulation. 2017 Sep 12;136(11):1049-1069. doi: 10.1161/CIRCULATIONAHA.117.028352. PMID 28893961
- [Background] Sammour Y, Krishnaswamy A, Kumar A, Puri R, Tarakji KG, Bazarbashi N, Harb S, Griffin B, Svensson L, Wazni O, Kapadia SR. Incidence, Predictors, and Implications of Permanent Pacemaker Requirement After Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2021 Jan 25;14(2):115-134. doi: 10.1016/j.jcin.2020.09.063. PMID 33478630
- [Background] Spears J, Al-Saiegh Y, Goldberg D, Manthey S, Goldberg S. TAVR: A Review of Current Practices and Considerations in Low-Risk Patients. J Interv Cardiol. 2020 Dec 24;2020:2582938. doi: 10.1155/2020/2582938. eCollection 2020. PMID 33447165